CLINICAL TRIAL: NCT03862729
Title: Risk Stratification and Minimally Invasive Surgery in Acute Intracerebral Hemorrhage Patients: a Prospective Multicenter Cohort Study (Risa-MIS-ICH Study)
Brief Title: Risk Stratification and Minimally Invasive Surgery in Acute ICH Patients
Acronym: Risa-MIS-ICH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Principal Investigator, Fuxin Lin, MD, First Affiliated Hospital of Fujian Medical University
Other Study IDs: GN-2018R002
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Spontaneous Intracerebral Hemorrhage
Keywords: Risk stratification; minimally invasive surgery; early-stage ICH patient; prospective cohort study
MeSH Terms: interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early minimally invasive surgery group: For patients in minimally invasive surgery group, intracranial hematoma will be removed by intraoperative stereotactic computer tomography-guided endoscopic surgery, or surgical aspiration followed by alteplase clot irrigation (1·0 mg every 8 h for up to nine doses). CTA will be performed before operation in all the patients for intraoperative navigation, and the minimally invasive surgery will be performed within 24 hours after intracerebral hemorrhage onset.
  Interventions: Procedure: Minimally invasive surgery
- conventional treatment group: Eligible patients not accepting early minimally invasive surgery are classified as the conventional treatment group. Conventional treatment includes medical treatment and conventional craniotomy. According to the intention-to-treat principle, patients treated by minimally invasive surgery beyond the 24 hours interval after ICH onset are also classified as conventional treatment group.
  Interventions: Procedure: conventional treatment

INTERVENTIONS:
Procedure: Minimally invasive surgery — Intracranial hematoma will be removed by intraoperative stereotactic computer tomography-guided endoscopic surgery, or surgical aspiration followed by alteplase clot irrigation (1·0 mg every 8 h for up to nine doses). CTA will be performed before operation in all the patients for intraoperative navigation, and the minimally invasive surgery will be performed within 24 hours after intracerebral hemorrhage onset.
  Groups: Early minimally invasive surgery group
Procedure: conventional treatment — Conventional treatment includes medical treatment and conventional craniotomy.
  Groups: conventional treatment group

SUMMARY:
The study consists of 2 parts: the first part is to conduct a multicenter retrospective analysis of more than 1000 acute ICH patients treated by conservative observation from 33 centers in China to create a predictive model of intracerebral hemorrhage growth based on clinical, blood, genetic, imaging, and pharmacological factors; the second part is to validate the efficacy of the minimally invasive surgery, including stereotactic thrombolysis and endoscopic surgery, in 300 eligible patients with high risk of hemorrhage growth according to the first part results in a prospective multicenter cohort study.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH) accounts for 2 million strokes worldwide per year and is the deadliest subtype of stroke with a 1-year mortality rate up to 50%. Given the high morbidity and mortality of this disease process, surgical options have been repeatedly evaluated in large multicenter randomized controlled trials that unfortunately have not demonstrated improved outcomes. Time to treatment is a factor that has been shown to carry enormous weight in the treatment of ischemic stroke but has not yet been demonstrated to play a role in hemorrhagic stroke. On the other hand, Intracerebral hemorrhage growth in early-stage is associated with the poor clinical outcome. Thus, investigators assume that minimally invasive surgery in early-stage ICH patients with high risk of hemorrhage growth may improve the long-term outcomes. In the first part, the investigators will review more than 1000 early-stage ICH patients from 33 centers within the last 5 years in China to create a predictive model of intracerebral hemorrhage growth based on clinical, blood, genetic, imaging, and pharmacological factors. The "early-stage" means 24 hours from symptom onset to baseline imaging. The "hemorrhage growth" is defined as an increase in intracerebral hemorrhage volume between baseline and repeat imaging of more than 6 mL or more than 33%. The second part is to validate the efficacy of the minimally invasive surgery in patients with high risk of hemorrhage growth according to the first part results in a prospective multicenter cohort study. Endoscopic surgery and stereotactic thrombolysis (150 patients) will be compared with conventional treatment (150 patients), including medical treatment and conventional craniotomy. Clinical data and laboratory data will be collected by electric case report form (CRF) and uploaded online by each neurosurgery center to form the prospective clinical database in First Affiliated Hospital of Fujian Medical University. This cohort follow-up study will be across a 3-year period with a 2 years interval of enrollment and 1 year follow up for each patient.

ELIGIBILITY:
1. Retrospective part

   Inclusion Criteria:
   * Emergent CT showed a spontaneous supratentorial intracerebral hemorrhage (patient with a small amount of intraventricular hemorrhage is eligible);
   * Patients should have undergone baseline CT scan within 48 hours after hemorrhage onset and repeated fewer than 48 hours after the baseline CT;
   * Patients without herniation.
   * Patients were treated by observation before hemorrhage growth (if happened).

   Exclusion Criteria:
   * Spontaneous intracerebral hemorrhage secondary to an underlying structural cause identified by brain imaging, (ie, vascular malformation, aneurysm, tumor);
   * The time from symptom onset to baseline imaging was not known in hours, clinical information or lab results was not enough to determine the growth of the hematoma or to perform statistical analysis;
   * Patients had accepted acute treatment that might have reduced intracerebral hemorrhage volume (ie, surgical evacuation, external ventricular drainage, lumbar puncture).
2. Prospective part

Inclusion Criteria:

* Emergent CT showed a spontaneous supratentorial intracerebral hemorrhage (patient with a small amount of intraventricular hemorrhage is eligible);
* Patients without herniation meet the clinical uncertainty principle as follows: the responsible neurosurgeon is uncertain about the benefits of surgery.
* Patients should have undergone baseline CT scan within 24 hours after hemorrhage onset; the volume of the hematoma is more than 20 ml and less than 100ml on the first CT scan.
* Patients with a Glasgow coma score of 5 or more.
* Informed consent, and willing to accept long-term follow-up.

Exclusion Criteria:

* Spontaneous intracerebral hemorrhage secondary to an underlying structural cause identified by brain imaging, (ie, vascular malformation, aneurysm, tumor);
* patients had a cerebellar hemorrhage or extension of a supratentorial hemorrhage into the brainstem;
* patients had severe pre-existing physical or mental disability or severe comorbidity that might interfere with the assessment of outcome.
* Severe coagulopathy, INR cannot be reversed to less than or equal to 1.5
* Patients during pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the retrospective part, at least 1000 conservatively treated acute ICH patients during the last 5 years from 31 Grade Ⅲ A level hospitals and 2 Grade Ⅱ A level hospitals distributed all over China will be enrolled. Patients should have undergone baseline CT scan within 24 hours after hemorrhage onset and repeated fewer than 48 hours. In the prospective part, at least 300 cute ICH patients with high risk of hemorrhage growth, according to the results of first part, from the same hospitals will be enrolled. All patients in this study should meet the inclusion and exclusion criteria. Informed written consent should be obtained from eligible adult patients or from the guardians of eligible pediatric patients. All patients in the prospective part of this study can withdraw at any time.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Severe disability or Death | 1 Year
  The prespecified primary endpoints are severe disability or death defined as Barthel Index ≤60 at 1 year after intracranial hemorrhage.

SECONDARY OUTCOMES:
All-cause mortality | 1 year
  Death caused by all the causes 1 year after enrollment.
Complications | 1 year
  Sever complications, including pulmonary embolism, adverse cardiac events, intracranial infection, re-hemorrhage, massive cerebral infarction and brain herniation happened within 1 month after hemorrhage onset.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available to other researchers after the main results of this study have been published.

REFERENCES:
- [Derived] Yao S, Gao Z, Fang W, Fu Y, Xue Q, Lai T, Shangguan H, Sun W, Lin Y, Lin F, Kang D. DPA714 PET Imaging Shows That Inflammation of the Choroid Plexus Is Active in Chronic-Phase Intracerebral Hemorrhage. Clin Nucl Med. 2024 Jan 1;49(1):56-65. doi: 10.1097/RLU.0000000000004948. Epub 2023 Nov 29. PMID 38054504
- [Derived] Li JB, Lin XR, Huang SN, He Q, Zheng Y, Li QX, Lin FX, Zhuo LY, Lin YX, Kang DZ, Ma K, Wang DL. High Plasma Fibrinogen Level Elevates the Risk of Cardiac Complications Following Spontaneous Intracerebral Hemorrhage. World Neurosurg. 2023 Dec;180:e774-e785. doi: 10.1016/j.wneu.2023.10.044. Epub 2023 Oct 13. PMID 37839573
- [Derived] Lin F, He Q, Zhuo L, Zhao M, Ye G, Gao Z, Huang W, Cai L, Wang F, Shangguan H, Fang W, Lin Y, Wang D, Kang D. A nomogram predictive model for long-term survival in spontaneous intracerebral hemorrhage patients without cerebral herniation at admission. Sci Rep. 2023 Feb 22;13(1):3126. doi: 10.1038/s41598-022-26176-0. PMID 36813798
- [Derived] Ye G, Huang S, Chen R, Zheng Y, Huang W, Gao Z, Cai L, Zhao M, Ma K, He Q, Lin F, Lin Y, Wang D, Fang W, Kang D, Wu X. Early Predictors of the Increase in Perihematomal Edema Volume After Intracerebral Hemorrhage: A Retrospective Analysis From the Risa-MIS-ICH Study. Front Neurol. 2021 Jul 27;12:700166. doi: 10.3389/fneur.2021.700166. eCollection 2021. PMID 34385972